CLINICAL TRIAL: NCT05684536
Title: Comparison of Liagure Safety in Thyroidectomy With Conventional Thyroidectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Imam Mohammad ibn Saud Islamic University (Other)
Responsible Party: Principal Investigator, mohammad bukhetan alharbi, associate professor, Imam Mohammad ibn Saud Islamic University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ligasure safety thyroidectomy
Record Dates: First submitted 2023-01-05; First posted 2023-01-13 (Actual); Last update posted 2023-01-13 (Actual); Status verified 2023-01

CONDITIONS: Ligature; Hemorrhage; Recurrent Laryngeal Nerve Injuries; Hypocalcemia
MeSH Terms: conditions — Hemorrhage; Recurrent Laryngeal Nerve Injuries; Hypocalcemia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ligasure throidectomy (Active Comparator): the vessel sealing device ( ligasure covidien ) which seals vessels by fusing the inner layers of the vessel wall, with dissection around ligament of berry and inferior thyroidal artery
  Interventions: Device: liagsure device
- conventional thyroidectomy (No Intervention): with dissection around ligament of berry and inferior thyroidal artery through ligation with vicryl and hemoclips

INTERVENTIONS:
Device: liagsure device — the vessel sealing device ( ligasure covidien ) which seals vessels by fusing the inner layers of the vessel wall, with dissection around ligament of berry and inferior thyroidal artery
  Arms: ligasure throidectomy

SUMMARY:
To compare intraoperative and postoperative complication rates in thyroidectomy between ligasure and traditional vascular ligation and clipping .

DETAILED DESCRIPTION:
Due to the high vascularity of the thyroid gland and the relatively tiny operative field, rigorous hemostasis is an essential requirement for successful thyroid surgery. Blood vessel ligation and/or ligation are the primary means of attaining hemostasis in thyroidectomy. New technologies have been developed, including a vessel sealing device (ligasure) that seals vessels by fusing the inner layers of the vessel wall with minimal amounts of thermal dispersion burning and tissue friction, thereby minimizing the occurrence of unintentional burns.

yet. It is unclear whether the heat conveyed by a ligature can harm the recurrent laryngeal nerve due to its proximity to the berry ligament.

thromosis of the inferior parathyroidal gland's supplying artery during dissection may result from alternative prospective delineation of the inferior thyroidal artery using ligasure for dissection.

The purpose of this study is to assess the safety and efficacy of ligasure with standard vascular ligation in open thyroid surgery.

ELIGIBILITY:
Inclusion Criteria:

Patient who will undergo lobectomy , subtotal thyroidectomy , total thyroidectomy at time of study

Any age

-

Exclusion Criteria:

* patient undergoing re-do surgery " completion thyroidectomy "

patient undergoing concomitant procedures as cervical lymphadenectomy or parathyroidectomy

Ages: 12 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-01-15 (Estimated); Primary Completion 2023-03-01 (Estimated); Study Completion 2023-04-01 (Estimated)

PRIMARY OUTCOMES:
Post-operative complications | Postoperatively from day of surgery until one week post operatively
  Including RLN palsy , hypocalcemia , hemorrhage wound infection